CLINICAL TRIAL: NCT03845062
Title: Contribution of Drug Induced Sleep Endoscopy in the Management of Pediatric Obstructive Sleep Apnea Hypopnea Syndrome
Brief Title: Contribution of Drug Induced Sleep Endoscopy of Pediatric Obstructive Sleep Apnea Hypopnea Syndrome
Acronym: ESSI
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0333
Record Dates: First submitted 2018-10-04; First posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2018-09

CONDITIONS: Obstructive Sleep Apnea Hypopnea Syndrome
Keywords: drug-induced sleep endoscopy; pediatric obstructive sleep apnea hypopnea syndrome; tongue base; epiglottis; occult laryngomalacia; lingual tonsillectomy; epiglottopexy; aryepiglottic folds division

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The role of drug-induced sleep endoscopy (DISE) in the management of obstructive sleep apnea hypopnea syndrome (OSAHS) is not precisely defined for children. The primary objective of this study was to describe the consequences of DISE in the therapeutic management for children with OSAHS. The secondary objectives were to analyze the correlation between the number of obstructive sites found during DISE, the value of apnea-hypopnea index (AHI), and the type of OSAHS.

DETAILED DESCRIPTION:
Retrospective single center study of 31 children (mean age: 5.5 ± 2.6 years) who benefited from DISE between 2015 and 2018 in the management of OSAHS. Modification of therapeutic management was noted. A correlation between the number of obstructive sites and the IAH on the one hand, and between the number of obstructive sites and the type of SAHOS on the other hand, was sought.

ELIGIBILITY:
Inclusion criteria:

- OSAHS confirmed by overnight sleep monitoring (respiratory polygraphy or overnight polysomnography)

Exclusion criteria:

- Lack of data

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with clinical obstructive sleep apnea hypopnea syndrome in University Health Center
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
sleep endoscopy | 1 day
  describe the modification of therapeutic management induced by sleep endoscopy

SECONDARY OUTCOMES:
Number of obstructive site during | 1 day
  retrospective data collection : Number of obstructive site during
value of apnea-hypopnea index | 1 day
  retrospective data collection : value of apnea-hypopnea index
type obstructive hypopnoea apnea syndrome of sleep | 1 day
  type obstructive hypopnoea apnea syndrome of sleep. Children facing craniofacial or neuromuscular disorders were rated in "Type III OSAHS". Obese children were rated in "Type II OSAHS". Others children were rated by default in "Type I OSAHS".

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Akkari, MD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France